CLINICAL TRIAL: NCT04083716
Title: A Phase 1, Open-Label, Randomized, 3-Way Crossover Study to Assess the Relative Bioavailability and Food Effect of ABI-H2158 in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability and Food Effect of ABI-H2158 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABI-H2158-102
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): ABI-H2158 Reference Formulation in a fasting state on Day 1 (Period 1), then ABI-H2158 Test Formulation in a fasting state on Day 8 (Period 2), then ABI-H2158 Test Formulation after a high-fat meal on Day 15 (Period 3)
  Interventions: Drug: ABI-H2158 Reference Formulation; Drug: ABI-H2158 Test Formulation
- Group 2 (Experimental): ABI-H2158 Test Formulation in a fasting state on Day 1 (Period 1), then ABI-H2158 Test Formulation after a high-fat meal on Day 8 (Period 2), then ABI-H2158 Reference Formulation in a fasting state on Day 15 (Period 3)
  Interventions: Drug: ABI-H2158 Reference Formulation; Drug: ABI-H2158 Test Formulation
- Group 3 (Experimental): ABI-H2158 Test Formulation after a high-fat meal on Day 1 (Period 1), then ABI-H2158 Reference Formulation in a fasting state on Day 8 (Period 2), then ABI-H2158 Test Formulation in a fasting state on Day 15 (Period 3)
  Interventions: Drug: ABI-H2158 Reference Formulation; Drug: ABI-H2158 Test Formulation

INTERVENTIONS:
Drug: ABI-H2158 Reference Formulation — ABI-H2158 tablets Reference Formulation
Drug: ABI-H2158 Test Formulation — ABI-H2158 tablets Test Formulation

SUMMARY:
This study is designed to assess the relative bioavailability of ABI-H2158 tablets (Test Formulation) compared to ABI-H2158 tablets (Reference Formulation). The effect of food on the pharmacokinetics of the Test Formulation will also be evaluated under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. No clinically significant abnormal findings on physical exam, medical history, or clinical laboratory results at screening.

Exclusion Criteria:

1. Positive test results for human immunodeficiency virus (HIV) or hepatitis B or C.
2. Treatment for drug or alcohol dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) of ABI-H2158: Relative Bioavailability and Food Effect | before dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dosing on Days 1, 8, and 15
Maximum observed plasma concentration (Cmax) of ABI-H2158: Relative Bioavailability and Food Effect | before dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dosing on Days 1, 8, and 15

CONTACTS AND LOCATIONS:
Overall Officials: Marc Evanchik, Study Director — Assembly Biosciences
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No